CLINICAL TRIAL: NCT00756743
Title: A Phase I Study To Evaluate The Safety, Tolerability, And Pharmacokinetics Of PF-04802540 After Multiple Oral Dose Administration To Healthy Adult Volunteers
Brief Title: Multiple Dose Safety Study of PF-04802540 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Taisho Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Taisho Pharmaceutical Co., Ltd.
Allocation: Randomized | Model: Crossover | Masking: Triple
Other Study IDs: B0911002
Record Dates: First submitted 2008-09-19; First posted 2008-09-22 (Estimated); Last update posted 2010-03-19 (Estimated); Status verified 2009-01

CONDITIONS: Healthy
Keywords: PF-04802540 multiple dose safety study

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- PF-04802540 (Experimental)
  Interventions: Drug: PF-04802540
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PF-04802540 — Multiple ascending doses for 10 days; planned doses include 5, 10 and 15 mg capsules q12 hours, doses may be adjusted based on accumulating data
  Arms: PF-04802540
Drug: Placebo — Placebo capsules q12 hours for 10 days
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, and pharmacokinetics of multiple ascending doses of PF-04802540 administered orally to healthy adult subjects.

DETAILED DESCRIPTION:
Evaluation of safety and pharmacokinetics

ELIGIBILITY:
Inclusion Criteria:

* Males or females of non-childbearing capacity aged 21 to 55 years inclusive at screening.
* Body mass index in the range of 18 to 30 kg/m2 and body weight>45 kg.
* Healthy as determined by the investigator on the basis of screening evaluation.

Exclusion Criteria:

* Use of prescription or nonprescription drugs
* Any condition possibly affecting drug absorption

Ages: 21 Years to 54 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2008-09; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Adverse events | 12 days
Safety assessments: vital signs, ECG, physical examination, laboratory tests | 12 days
Pharmacokinetics | 12 days

SECONDARY OUTCOMES:
No secondary outcomes measures. | Timeframe N/A

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Singapore, Singapore

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B0911002&StudyName=Multiple%20Dose%20Safety%20Study%20of%20PF-04802540%20in%20Healthy%20Volunteers%0A%0A